CLINICAL TRIAL: NCT05646511
Title: A Multicenter Randomized Phase III Study of Short-term Radiotherapy Plus CAPOX and Short-term Radiotherapy Plus CAPOXIRI as Preoperative Treatment for Locally Advanced Rectal Cancer
Brief Title: TNT of SCRT+CAPOX vs SCRT+CAPOXIRI for Locally Advanced Rectal Cancer
Acronym: ENSEMBLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Takayuki Yoshino, MD., PhD Head of Department of Gastroenterology and Gastrointestinal Oncology, National Cancer Center Hospital East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2022001; jRCTs031220342 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Radiation; CAPOXIRI; CAPOX; Rectal cancer; Total neoadjuvant therapy; Rectal Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Capecitabine; Oxaliplatin; Irinotecan; Antineoplastic Agents; Chemotherapy; Non-operative management; Surgery; MRI; Restaging; QOL; Organ preservation; TNT
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Intervention Model Description: standard arm: 5x5Gy - - 12 wks CAPOX- - restaging - - surgery or non-operative management experimental arm: 5x5Gy - - 12 wks CAPOXIRI - - restaging - - surgery or non-operative management
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm SCRT+CAPOX (Active Comparator): The standard-of-care group receives short-course radiation therapy (5 × 5 Gy) followed by six cycles of CAPOX (capecitabine 1000 mg/m2 orally twice daily on days 1-14, oxaliplatin 130 mg/m2 intravenously on day 1, q3wks).
  Interventions: Radiation: SCRT; Drug: CAPOX
- Experimental arm SCRT+CAPOXIRI (Experimental): The standard-of-care group receives short-course radiation therapy (5 × 5 Gy) followed by six cycles of CAPOXIRI (capecitabine 800 mg/m2 orally twice daily on days 1-14, oxaliplatin 130 mg/m2 intravenously on day 1, and irinotecan 150 mg/m2 intravenously on day 1*, q3wks).
  Interventions: Radiation: SCRT; Drug: CAPOXIRI

INTERVENTIONS:
Radiation: SCRT — 5x5 Gy: 25 Gy
  Other Names: Active Comparator & Experimental
Drug: CAPOX — Six cycles of CAPOX capecitabine 1000 mg/m2 orally twice daily on days 1-14, oxaliplatin 130 mg/m2 intravenously on day 1, every 3 weeks
  Other Names: Active Comparator
  Arms: Control arm SCRT+CAPOX
Drug: CAPOXIRI — Six cycles of CAPOXIRI capecitabine 800 mg/m2 orally twice daily on days 1-14, oxaliplatin 130 mg/m2 intravenously on day 1 and irinotecan 150 mg/m2 intravenously on day 1, every 3 weeks
  Other Names: Experimental
  Arms: Experimental arm SCRT+CAPOXIRI

SUMMARY:
This trial is a multicenter randomized Phase III study to verify the superiority of short-course preoperative radiation (SCRT) and CAPOXIRI over SCRT and CAPOX as preoperative treatments for locally advanced rectal cancer.

DETAILED DESCRIPTION:
Total neoadjuvant therapy (TNT) for locally advanced rectal cancer (LARC) has the promise, which means non-operative management (NOM) enable more patients (pts) with a complete clinical response (cCR) or near-complete clinical responses (nCR) after TNT to avoid subsequent radical surgery, with potentially maintaining anorectal function and quality of life (QoL). Recently, PRODIGE-23 trial demonstrated that triplet regimen (Irinotecan, oxaliplatin and fluoropyrimidine) before preoperative chemoradiotherapy (CRT) significantly improved outcomes compared with CRT. However, there has been no prospective study comparing consolidation triplet with doublet regimens following short course radiotherapy (SCRT). The aim of this randomized phase III trial is to test superiority of consolidation irinotecan, capecitabine and oxaliplatin (CAPOXIRI) vs. capecitabine and oxaliplatin (CAPOX) following SCRT as TNT in pts with LARC.

Pts in both groups will be re-staged after completing TNT before radical surgery according to the Memorial Sloan Kettering Regression Schema; pts with incomplete response (iCR) will undergo total mesorectal excision (TME), cCR pts will receive NOM, and nCR pts will undergo TME or NOM by a physician discretion under the recommendation of blind assessment by the designated NOM central committee. Pts will be followed by CT, MRI, colonoscopy and liquid biopsy every 4 months for 2 years, and every 6 months thereafter up to 5 years.

To detect a decrease in 3-year cumulative probability of organ preservation-adapted Disease free survival (DFS) from 75.0% to 81.7%, corresponding to a target hazard ratio of 0·70, a total of 608 pts (196 events) would achieve 70% power at a two-sided α significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. The content of this research was fully explained, and written informed consent was obtained from the subject.
2. Histologically confirmed rectal adenocarcinoma.
3. Radical resection is clinically possible without any distant metastases on imaging studies.
4. Age of 18 years or older on the date of consent acquisition.
5. Eastern Cooperative Oncology Group (ECOG) PS 0-1 (PS 0 if aged 70 years or older on consent acquisition date).
6. Inferior margin of the tumor is within 12 cm of the AV.
7. No prior tumor treatment.
8. No history of radiation therapy to the pelvis, including treatment for other cancer types.
9. Cases with cT3-4N0M0*or T1-4N1-2M0 based on Union Internationale Contre le Cancer (UICC) 8th edition.

   (*5 cm< AV ≤ 10 cm, T3a/bN0M0, extramural venous invasion (EMVI) -, mesorectal fascia (MRF) clear and 10 cm < AV ≤ 12 cm, T3a/bN0-1M0, EMVI-, MRF clear are eligible only for those who refused surgery)
10. UGT1A1 is wild-type or single heterozygous.
11. Criteria for major organ function within 28 days prior to enrollment. If there are multiple test results within this period, the most recent one will be used, and blood transfusions and hematopoietic factor preparations will not be administered within 14 days before the test date for measurements before registration.

    1. Neutrophil count: ≥1,500/mm3
    2. Platelet count: ≥10.0×10 4/mm3
    3. Hemoglobin concentration: ≥9.0 g/dL
    4. Total bilirubin: ≤2.0 mg/dL
    5. Aspartate transaminase (AST): ≤100 IU/L or less
    6. Alanine transaminase (ALT): ≤100 IU/L or less
    7. Serum creatinine: Creatinine clearance ≥30 mL/min (by Cockcroft & Gault formula)

Exclusion Criteria:

1. Extensive surgery (excluding colostomy and central venous port construction) within 4 weeks before starting protocol treatment.
2. Complications or history of severe lung disease (such as interstitial pneumonia, pulmonary fibrosis, and severe emphysema).
3. Colonic stent in place.
4. Contraindications for MRI such as cardiac pacemakers.
5. Serious comorbidities (such as heart failure, renal failure, liver failure, intestinal paralysis, intestinal obstruction, uncontrolled diabetes, and active inflammatory bowel disease).
6. Patients with multiple active cancers (simultaneous multiple cancers or metachronous multiple cancers with a disease-free interval of 5 years or less). However, carcinoma in situ or lesions equivalent to intramucosal carcinoma, which can be cured by local treatment, are not treated as active multiple cancers.
7. Pregnant women, lactating women, positive pregnancy test, or unwillingness to use contraception.
8. Hepatitis B surface (HBs) antigen positive or hepatitis C virus (HCV) antibody-positive. However, HCV-RNA-negative can be registered.
9. Have human immunodeficiency virus (HIV) infection.
10. MSI-high (MSI-H) or defective mismatch repair (dMMR) is known.
11. Unwilling to donate specimens for "Research on gene profiling and clinical significance using clinical specimens from cancer patients" for whole-genome analysis based on the "Action Plan for Whole-Genome Analysis, etc." (CONDUCTOR study).
12. Any other patients the principal investigator or co-investigator deems inappropriate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Organ-preservation adapted DFS | Up to 3 years. It is defined as the period from the allocation date to the earliest of the following events.
  The investigators use the definition of organ-preservation adopted DFS proposed in the international consensus statement for preoperative treatment (75). It is defined as the period from the date of allocation to the earliest of the following events.
  1. Surgery difficult due to local progression or study subject unfit for surgery
  2. R2 resection of primary tumor ( not including Circumferential resection margin (CRM) positive )
  3. Local recurrence after R0/1 resection of primary tumor
  4. Local regrowth for which Salvage surgery is not possible during NOM
  5. Appearance of distant metastases
  6. Occurrence of second primary colorectal cancer
  7. Development of second primary other cancers
  8. Death (treatment-related death, death from the same cancer, death from a different type of cancer, non-cancer-related death)

SECONDARY OUTCOMES:
cCR rate | 1-3 weeks (Days 7-21) from the completion of preoperative chemotherapy or the date of discontinuation.
  The investigators will use the Memorial Sloan Kettering Regression Schema, which is the cCR standard for TNT clinical trials conducted mainly in the United States.
  For judgment, a gastrointestinal endoscopist, a pathological diagnostician, and a gastrointestinal surgeon discuss and comprehensively judge.
Clinical response (cCR+near CR [nCR]) rate | Within 1-3 weeks (Days 7-21) from the completion of preoperative chemotherapy or the date of discontinuation.
  The investigators will use the Memorial Sloan Kettering Regression Schema, which is the cCR standard for TNT clinical trials conducted mainly in the United States.
  For judgment, a gastrointestinal endoscopist, a pathological diagnostician, and a gastrointestinal surgeon discuss and comprehensively judge.
Proportion of NOM selection | 3-6 weeks (Days 21-42) from the completion of preoperative chemotherapy or the date of discontinuation.
  The proportion of the number of research subjects for whom NOM was selected at the time of re-evaluation to the analysis population as the numerator. Study subjects who died of any cause before the re-evaluation decision date will be treated as "no complete resection" and included in the denominator but not the numerator.
Recurrence type and recurrence rate | 3 years (up to 5 years)
  The recurrence site is classified into local recurrence, distant recurrence, and unknown, and is defined as "recurrence type". Select multiple categories if recurrence is observed at multiple sites at the time of the first recurrence.
Distant metastases free survival (DMFS) | 3 years (up to 5 years)
  The period from the date of allocation to the date of determination of distant metastasis or the date of death due to any cause, whichever is earlier. An event that corresponds to any of the following is defined as a DMFS event.
  1. Distant metastasis
  2. Death (treatment-related death, death from the same cancer, death from a different type of cancer, non-cancer-related death)
Local recurrence-free survival (LRFS) | 3 years (up to 5 years)
  The period from the date of allocation to the date of local recurrence or the date of death due to any cause, whichever is earlier. An event that corresponds to any of the following is defined as an LRFS event.
  1. Local recurrence
  2. Death (treatment-related death, death from the same cancer, death from a different type of cancer, non-cancer-related death)
Overall survival (OS) | 3 years (up to 5 years)
  From the date of allocation to the date of death due to any cause. Based on " Protocol 8.2.17 Confirmation of outcome and confirmation of recurrence after protocol treatment", the confirmation of survival should be recorded in the medical record, etc.). Patients with no follow-up will be censored on the date of final confirmation of survival.
TME-free survival | 3 years (up to 5 years)
  As the earliest of the date of definitive TME at reevaluation, the date of TME at local recurrence (excluding local excision), and the date of death from any cause. An event corresponding to any of the following is defined as a TME free survival event.
  1. TME when electing surgery at reevaluation
  2. TME with salvageable local regrowth in NOM
  3. Death (treatment-related death, death from the same cancer, death from a different type of cancer, non-cancer-related death)
TME-free DFS | 3 years (up to 5 years)
  With the date of assignment as the starting date, the date on which radical TME was performed at reevaluation, the date on which TME was performed at the time of local recurrence (excluding local excision), and Organ-preservation adopted DFS defined in Protocol 12.2.1. The period up to the earliest of the event occurrence dates. An event that corresponds to any of the following is defined as an event of TME-free disease-free survival.
  1. TME when electing surgery at reevaluation
  2. TME with salvageable local regrowth in NOM
  3. Organ preservation - adopted DFS defined in Protocol 12.2.1. is not applicable because TME is implemented)
Protocol treatment completion rate | Immediately after the completion of preoperative chemotherapy or the date of discontinuation.
  The analysis population who completed protocol treatment.
Relative dose intensity (RDI) | Immediately after the completion of preoperative chemotherapy or the date of discontinuation.
  RDI is calculated for each case, each cycle, and each drug (capecitabine, oxaliplatin, irinotecan) in the analysis target population. The actual number of cycle days refers to the number of days from the start of the corresponding course to the start date of the next course, but the actual number of cycle days in the final course is the number of days from the start date of the last course to the actual day of administration of capecitabine + 6 days. defined as RDI (%) = (Actual Dose/Prescribed Dose) x (21/Actual Cycle Days) x 100
QOL assessment (LARS score, EORTC QLQ-C30, and SF-36) | 3 years
  Using a quality of life questionnaire to assess the following items: LARS score, EORTC QLQ-C30, SF-36
Incidence of preoperative treatment-related adverse events | Immediately after the completion of preoperative chemotherapy or the date of discontinuation.
  Incidence of preoperative treatment-related adverse events determined by CTCAE ver5.0
Pathological complete response (pCR) rate in the surgical subgroup | Immediately after the evaluation of the histopathological findings after surgery
  Pathological response evaluation will be performed on the surgical specimens of the subgroup that underwent surgical resection in the protocol treatment.
  Histopathological evaluation of antitumor efficacy is based on the American Joint Committee on Cancer (AJCC) evaluation method. pCR is defined as no viable tumor cells not only in the primary tumor but also in the regional lymph nodes (ypT0N0).
  Percentage of study subjects judged to be pCR in the analysis population.
Radical resection rate in the surgical subgroup | 3 years (up to 5 years)
  Proportion of study participants who underwent a complete resection (confirmed postoperative pathological R0) in the analyzed population in the surgical resection subgroup in protocol treatment. Study subjects who died of any cause prior to the date of surgery were treated as "no complete resection" and included in the denominator but not the numerator.
Local recurrence-free survival (LRFS) in the surgical subgroup | 3 years (up to 5 years)
  In the subgroup that underwent surgical resection in protocol treatment, the period from the date of surgery to the date of local recurrence or the date of death from any cause, whichever comes first.
Surgery-related adverse event rate determined by Clavien-Dindo classification v2.0 in the surgical subgroup | For early (within 30 days) and late (31-90 days) postoperative adverse events after the end of surgical therapy
  For early (within 30 days) and late (31-90 days) postoperative adverse events after the end of surgical therapy, the worst grade according to the Clavien-Dindo classification v2.0 is calculated.
Local re-enlargement rate in the NOM subgroup | 3 years (up to 5 years)
  Proportion of study subjects with local regrowth in the analysis population in the subgroups that underwent NOM.
Time for local regrowth in the NOM subgroup | 3 years (up to 5 years)
  In the subgroup that underwent NOM, the date of NOM determination is the starting date, and the period from the date of local regrowth to the date of death from any cause, whichever is earlier.
Proportion of salvage surgery in local re-enlargement cases in the NOM subgroup | 3 years (up to 5 years)
  In the NOM subgroup, the proportion of study subjects with local regrowth and salvage surgery in the analysis population.
Time until salvage surgery in the NOM subgroup | 3 years (up to 5 years)
  In the NOM subgroup, the time to the date of salvage surgery at the time of local regrowth or the date of death from any cause, whichever is earliest.
Surgery-related adverse event rate determined by Clavien-Dindo classification v2.0 in salvage surgery cases in the NOM subgroup | For early (within 30 days) and late (31-90 days) postoperative adverse events after the end of surgical therapy
  In the subgroup that underwent NOM, among the population to be analyzed, in cases where local regrowth was performed and salvage surgery was performed, early (within 30 days) and late (31-90 days) postoperative adverse events after the end of surgical therapy , find the worst grade by Clavien-Dindo classification v2.0.
Proportion of radical resection in salvage surgery cases in the NOM subgroup | 3 years (up to 5 years)
  Proportion of study subjects with local regrowth and radical salvage surgery in the analyzed population in the NOM subgroup.

OTHER OUTCOMES:
liquid biopsy | 3 years (up to 5 years)
  Analysis using liquid biopsy will be performed to identify biomarkers that predict therapeutic effects by performing blood genome profiling.
Artificial Intelligence (AI) (deep learning) analysis | 3 years (up to 5 years)
  Using multiple algorithms, in addition to colonoscopy and pelvic MRI images at each point, clinicopathological features, various biomarkers, and QOL will be utilized to estimate the optimal treatment method for individual research subjects

CONTACTS AND LOCATIONS:
Locations (34):
- Japan (34):
  - National Cancer Center Hospital East, Chiba
  - Ehime Prefectural Central Hospital, Ehime
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Gifu University Hospital, Gifu
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - St. Marianna University Hospital, Kawasaki
  - University of Occupational and Environmental Health Hospital, Kitakyushu
  - Kochi Medical School Hospital, Kochi
  - Kumamoto University Hospital, Kumamoto
  - Kyoto Prefectural University of Medicine, Kyoto
  - Nagoya University Hospital, Nagoya
  - Ohara Memorial Kurashiki Central Medical Organization Kurashiki Central Hospital, Okayama
  - Okayama University Hospital, Okayama
  - Kansai Medical University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - National Hospital Organization Osaka Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka Prefectural Hospital Organization Osaka Acute and General Medical Center, Osaka
  - Osaka University Hospital, Osaka
  - Kitasato University Hospital, Sagamihara
  - Sapporo Medical University Hospital, Sapporo
  - Keio University Hospital, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Hospital Organization Tokyo Metropolitan Komagome Hospital, Tokyo
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama
  - Yokohama City University Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Federation of National Public Service Personnel Mutual Aid Associations Yokosuka Mutual Aid Hospital, Yokosuka

IPD SHARING:
Plan to Share IPD: Yes
A part of the omics analysis data obtained in the analysis of this study may be disclosed through public databases such as the "Human Database" operated by National Bioscience Database Center (NBDC) in Japan Science and Technology Agency (JST). When registering data, re-anonymization will be provided to strengthen the protections of personal information. At the time of NBDC registration, we will comply with the "NBDC Guidelines for Human Data Sharing" and "NBDC Security Guidelines for Human Data(for Data Providers)" .

REFERENCES:
- [Background] Watanabe J, Kagawa Y, Chida K, Ando K, Kotani D, Oba K, Bando H, Hojo H, Shimamoto S, Sakashita S et al: Phase III trial of short-course radiotherapy followed by CAPOXIRI versus CAPOX in locally advanced rectal cancer: the ENSEMBLE trial. ESMO Gastrointestinal Oncology 2023, 1:9-14.
- [Background] Kagawa Y, Smith JJ, Fokas E, Watanabe J, Cercek A, Greten FR, Bando H, Shi Q, Garcia-Aguilar J, Romesser PB, Horvat N, Sanoff H, Hall W, Kato T, Rodel C, Dasari A, Yoshino T. Future direction of total neoadjuvant therapy for locally advanced rectal cancer. Nat Rev Gastroenterol Hepatol. 2024 Jun;21(6):444-455. doi: 10.1038/s41575-024-00900-9. Epub 2024 Mar 14. PMID 38485756
- [Background] Scott AJ, Kennedy EB, Berlin J, Brown G, Chalabi M, Cho MT, Cusnir M, Dorth J, George M, Kachnic LA, Kennecke HF, Loree JM, Morris VK, Perez RO, Smith JJ, Strickland MR, Gholami S. Management of Locally Advanced Rectal Cancer: ASCO Guideline. J Clin Oncol. 2024 Oct;42(28):3355-3375. doi: 10.1200/JCO.24.01160. Epub 2024 Aug 8. PMID 39116386
- [Background] Kagawa Y, Watanabe J, Uemura M, Ando K, Inoue A, Oba K, Takemasa I, Oki E. Short-term outcomes of a prospective multicenter phase II trial of total neoadjuvant therapy for locally advanced rectal cancer in Japan (ENSEMBLE-1). Ann Gastroenterol Surg. 2023 Jul 11;7(6):968-976. doi: 10.1002/ags3.12715. eCollection 2023 Nov. PMID 37927927
- [Background] Kagawa Y, Ando K, Uemura M, Watanabe J, Oba K, Emi Y, Matsuhashi N, Izawa N, Muto O, Kinjo T, Takemasa I, Oki E. Phase II study of long-course chemoradiotherapy followed by consolidation chemotherapy as total neoadjuvant therapy in locally advanced rectal cancer in Japan: ENSEMBLE-2. Ann Gastroenterol Surg. 2024 Aug 3;8(6):1067-1075. doi: 10.1002/ags3.12848. eCollection 2024 Nov. PMID 39502728